CLINICAL TRIAL: NCT04253275
Title: Identification of Biomarkers in Ischemic Stroke - Clinical Trial
Acronym: IBIS-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBIS-CT (29BRC19.0268)
Record Dates: First submitted 2020-01-07; First posted 2020-02-05 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ischemic stroke patients (Other): Patients with ischemic stroke diagnosed on clinical presentation and cerebral imaging
  Interventions: Genetic: blood samples
- hemorragic stroke patients (Other): Patients with hemorragic stroke diagnosed on clinical presentation and cerebral imaging
  Interventions: Genetic: blood samples
- healthy controls (Other): Stroke-free
  Interventions: Genetic: blood samples; Diagnostic Test: MRI without injection

INTERVENTIONS:
Genetic: blood samples — Blood samples will be taken at inclusion, 12h, 24h, 48h, 7d, 3m and 1y for patients ; at inclusion, 3m and 1y for controls.
  Microvesicles samples will be taken at inclusion, 7d and 3M ; at inclusion and 3M for controls.
Diagnostic Test: MRI without injection — MRI at inclusion for controls
  Arms: healthy controls

SUMMARY:
The objective of the study is to determine RNA blood biomarker based on 9 genes already identified in experimental studies, whose expression would be significantly increased in patient with ischemic stroke compared to controls.

DETAILED DESCRIPTION:
This is a monocentric study. It's a case-control study with case being first-ever ischemic stroke and controls being healthy (stroke free) subject patients paired for age, sex and cardiovascular risk or hemorrhagic stroke paired for age and sex.

Patients are followed for one year. Blood samples will be taken at inclusion, 12h, 24h, 48h, 7d, 3m and 1y. Microvesicles samples will be taken at inclusion, 7d and 3M.

ELIGIBILITY:
Inclusion Criteria:

* For ischemic stroke :
* Age > 18-year-old
* Ischemic stroke diagnosed on clinical presentation and cerebral imaging (CT or MRI imaging)
* Inclusion inferior to 6 hours from stroke onset
* Initial NIHSS score > 0 at the time of clinical examination
* Patients with multimodal imaging either through MRI or CT perfusion and supra-aortic vessels and intra-cerebral vessels (Willis circle) imaging <0
* Procedure of signed consent in situation of emergency : consent of the patient if he has the possibility to sign or his representative if he is present
* For hemorragic stroke :
* Age > 18 year-old
* Hemorrhagic stroke diagnosed on clinical presentation and cerebral imaging (CT or MRI imaging)
* Inclusion inferior to 6 hours from stroke onset
* Initial NIHSS score > 0 at the time of clinical examination
* Hemorrhagic patients are paired for age and sex with ischemic patients
* Procedure of signed consent in situation of emergency : consent of the patient if he has the possibility to sign or his representative if he is present

For healthy controls :

* Age > 18 year-old
* Stroke-free standardized questionnaire
* Initial NIHSS score = 0
* Rankin score = 0
* High risk cardiovascular subjects
* Controls are paired for age, sex and cardiovascular risk measured by a score (European Heart Score) with ischemic patients

Exclusion Criteria:

* Not affiliated to social security
* Patient under legal protection or deprived of liberty by a judicial or administrative decision
* Patient whose follow-up will be impossible
* Prior stroke

GROUP FOR ISCHEMIC STROKE :

- Patients with TIA and a negative cerebral CT or MRI

GROUP FOR HEMORRAGIC STROKE :

* Cerebral hemorrhage related to subarachnoid hemorrhage
* Post-traumatic hemorrhage
* Hemorrhagic transformation in patients with ischemic stroke

GROUP FOR HEALTHY CONTROLS :

- Contraindication MRI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Expression (measured in log2) of each 9 targeted genes identified less than 6 hours after inclusion | 6 hours after inclusion
  Each targeted genes will be measured by quantitative reverse transcription Polymerase Chain Reaction (rt-PCR)

SECONDARY OUTCOMES:
RNA level expression across time according growth of infarction measured at inclusion and at 3 months | inclusion and 3 months
  Each targeted genes will be measured by quantitative rt-PCR
RNA level expression across time according Rankin scale at three months dichotomized in good (≤ 2) and bad prognosis (> 3). | at 3 months
  Each targeted genes will be measured by quantitative rt-PCR
Targeted RNA level expression according mechanism of ischemic stroke | at 3 months
  Each targeted RNA level expression of targeted genes will be measured by quantitative rt-PCR
Target RNA level expression in the saliva | at inclusion
  For 3 participants, one of each arm, a saliva sample will be collected at inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Serge TIMSIT, Pr, Principal Investigator — serge.timsit@chu-brest.fr
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.